CLINICAL TRIAL: NCT00944268
Title: Clinical Study Phase III, Multicenter, Prospective, Open to Evaluate the Efficacy and Tolerability of the Combination Use of Passiflora Incarnata L, Crataegus Oxyacantha and Salix Alba L in Mild and Moderate Anxiety
Brief Title: Efficacy and Tolerability Study to Treat Mild and Moderate Anxiety
Acronym: E01ATCAL0308
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ativus Farmaceutica Ltda (Industry)
Responsible Party: Olinto Mascarenhas Marques, ATIVUS FARMACÊUTICA LTDA
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: E01-AT-CAL-03-08
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2009-07-24 (Estimated); Status verified 2009-07

CONDITIONS: Anxiety; Efficacy; Tolerability
Keywords: Passiflora, Crataegus and Salix; Mild and Moderate anxiety; Tablet; To evaluate the efficacy and tolerability of the combination
MeSH Terms: conditions — Anxiety Disorders; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liquid and solid (Experimental)
  Interventions: Drug: Passiflora, Crataegus e Salix

INTERVENTIONS:
Drug: Passiflora, Crataegus e Salix — Comparison of different pharmaceutics forms of drug

SUMMARY:
To evaluate the efficacy and tolerability of the combination use of Passiflora incarnata L, Crataegus oxyacantha and Salix alba L in mild and moderate anxiety.

Clinical study phase III, multicenter, prospective, open.

Patients will be included in sufficient quantity to achieve the minimum number of 124 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who achieve scores between 18 and 29 points in the Hamilton Scale for Anxiety;
* Individuals of any ethnic group male and female, aged above 18 years;
* Consent of the subject of research (a consent form signed).

Exclusion Criteria:

* Patients with known hypersensitivity to any components of the formula;
* Pregnant women and nursing mothers;
* Patients with endogenous depression, schizophrenia, suicidal tendency;
* Patients with heart disease unabated, unabated kidney, liver and lung unabated unabated, at the discretion of the investigator;
* Addiction to drugs, including alcohol, at the discretion of the investigator;
* Patients who are using any medication that could interfere with the effect of the drug under study;
* Impossibility of compliance to the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2009-09; Primary Completion 2009-12 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Scales | 30 days

SECONDARY OUTCOMES:
Safety evaluation by adverse events relate. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Elie Fiss, Principal Investigator — Faculdade de Medicina do ABC
Locations (1):
- Faculdade de Medicina do ABC, Santo André, São Paulo, Brazil